CLINICAL TRIAL: NCT06710782
Title: A Comparative Study Between Transcutaneous Pulsed Radiofrequency Application Plus Genicular Nerve Block Versus Intra-Articular Hyaluronic Acid Injection for Management of Chronic Pain in Knee Osteo-arthritis: A Prospective Randomized Controlled Study.
Brief Title: Transcutaneous Pulsed Radiofrequency Application Plus Genicular Nerve Block Versus Intraarticular Hyaluronic Acid Injection for Management of Chronic Pain in Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Omar Hashem Mohammed, Resident of Anesthesiology,Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS262/7/23
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Transcutaneous; Pulsed Radiofrequency; Genicular Nerve Block; Intraarticular; Hyaluronic Acid; Chronic Pain; Knee Osteoarthritis
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic Acid group (Experimental): Patients underwent intra-articular hyaluronic acid injection.
  Interventions: Drug: Hyaluronic acid
- Transcutaneous pulsed radiofrequency group (Experimental): Patients underwent transcutaneous pulsed radiofrequency application plus genicular nerve block.
  Interventions: Device: Transcutaneous pulsed radiofrequency

INTERVENTIONS:
Drug: Hyaluronic acid — Patients underwent intra-articular hyaluronic acid injection.
  Arms: Hyaluronic Acid group
Device: Transcutaneous pulsed radiofrequency — Patients underwent transcutaneous pulsed radiofrequency application plus genicular nerve block.
  Arms: Transcutaneous pulsed radiofrequency group

SUMMARY:
The aim of the present study is to compare the analgesic efficacy of combined transcutaneous pulsed radiofrequency plus genicular nerve block with bupivacaine plus corticosteroid versus intraarticular Hyaluronic acid injections, in terms of clinical and functional parameters, in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Total knee arthroplasty is commonly used as a surgical option for the treatment of symptomatic knee osteoarthritis to relieve pain and improve function, although it is associated with increased perioperative morbidity and mortality, particularly in older patients with co morbidities. Despite high success rates after total knee arthroplasty , a significant number of patients report suffering from postoperative pain, which can be worse than reported preoperative pain.

As an alternative approach, radiofrequency treatment modalities on the knee joint have been used to reduce knee pain due to osteoarthritis. Genicular nerve block (GNB) is a recently developed therapeutic option for knee osteoarthritis. that targets the three sensory nerves of the knee: superior lateral, superior medial and inferior medial genicular nerve, to inhibit pain transmission to the central nervous system.

Early osteoarthritis. treatment combines non pharmacological techniques with oral pharmacological therapies, intraarticular injections (IAI) of hyaluronic acid (HA), corticosteroid with local anesthetic or platelet-rich plasma (PRP) are used in progressive or very symptomatic stage. Intraarticular injections (IAI) is considered one of first-line treatments in recent studies as it is effective in decreasing pain and safer than oral pharmacological therapies.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 40 years.
* Both sexes
* American Society of Anesthesiologists (ASA)physical status I and II.
* Patients radiologically proven symptomatic knee joint osteoarthritis not responding to medical treatment.
* Patients with knee pain of moderate or greater intensity on most or all days for ≥ 3 months, showing significant radiological osteoarthritis (Kellgren-Lawrence grade 1 to 3).

Radiological severity was assessed using the Kellgrenand Lawrence global scale as follow: Grade 0; means absence of radiological finding; grade 1: suspected narrowing of joint space; grade 2 refers to osteophytes and possible narrowing; grade 3 is defined as multiple os-teophytes, definite narrowing of joint space and grade 4 comprises large osteophytes, marked narrowing of joint space.

Exclusion Criteria:

* Patient refusal.
* Patients who show improvement on medical treatment, patients on an oral, topical, or intra-articular steroid during the 4 weeks before the study; patients with an oral, topical, or suppository non-steroidal anti-inflammatory drugs within 2 weeks before the study.
* Patients having secondary knee osteoarthritis.
* Patients with severe osteoarthritis.(K/L grade >3) in a location other than the knee joint.
* Patients with rheumatoid arthritis.
* Patients with joint replacement surgery in either knee and/or a hip.
* Patients with meniscal tear, ligament injury, bursitis, and popliteal cyst and blood investigations suggestive of any infection.
* Morbid obese patients (body mass index (BMI) of >40 kg/m2)
* Infection at site of injection.
* Bleeding diathesis and coagulopathy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Degree of pain | 3 month after injection
  Assessment of pain severity by visual analog scale (VAS) at the baseline (before injection), 1month and 3month, intervals after injection.
  The visual analog scale (VAS) score it has 10-cm scale that represents a continuum between "0 = no pain" and "10 = worst pain."

SECONDARY OUTCOMES:
Functional status | 3 month after injection
  Functional status and daily activity via the western ontario and mcmaster universities osteoartheritis index (WOMAC) score before one month and three monthes after injection.
  The WOMAC consists of three subscales: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores represent worse pain, stiffness, and functional limitations.
Daily activity | 3 month after injection
  Daily activity via the western ontario and mcmaster universities osteoartheritis index (WOMAC) score before one month and three monthes after injection.
  The WOMAC consists of three subscales: pain (five questions), stiffness (two questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores represent worse pain, stiffness, and functional limitations.
Analgesic requirement | 3 month after injection
  Analgesic requirement (Dose and frequency of oral acetaminophen intake) for post injection pain if visual analogue scale (VAS) more than 3.
  Visual Analogue Scale (VAS) used as an effective tool to detect intensity of pain was recorded;"0" represents no pain,"10" worst pain, "1-3" mild pain,"4-6 " moderate pain and" 7-10 " severe pain
Adverse events | 3 month after injection
  Adverse events were recorded such as toxicity of local anesthetic drug occur, the research was stopped and was cleared to ehtical committees.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data was available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data was available upon a reasonable request from the corresponding author.